CLINICAL TRIAL: NCT01614106
Title: Project RETAIN: Providing Integrated Care for HIV-Infected Crack Cocaine Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Emory University (Other); University of Miami (Other); The Village South (Other); Grady Health System (Other); Jackson Health System (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa Metsch, Stephen Smith Professor and Chair of Sociomedical Sciences Department, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAK0606; R01DA032098 (NIH)
Record Dates: First submitted 2012-03-14; First posted 2012-06-07 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: HIV; AIDS; Substance Abuse
Keywords: HIV/AIDS; Drug Users; Crack-Cocaine Use; HIV Primary Care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Retention Clinic will incorporate HIV primary care and mental health services with on-site substance abuse treatment and patient navigation. The central components will include: Primary HIV Care; Mental Health Services; Skill-building; and On-Site substance abuse treatment (including Motivational Enhancement Therapy and Cognitive Behavioral Therapy).
  Interventions: Behavioral: Retention Clinic
- Treatment as Usual (TAU) (No Intervention): The treatment as usual (TAU) group condition will represent standard of care at both of the participating clinics. Standard of care at both clinics includes primary HIV care, the provision of mental health services, and the assignment of a clinic case manager. These case managers meet with patients when they first come to clinic and then meet with them as needed and typically offer substance-using patients a referral to substance abuse treatment in the community as needed. Case managers usually do not follow up to determine the uptake of these referrals.

INTERVENTIONS:
Behavioral: Retention Clinic — The central components of the Retention Clinic will include: Primary HIV Care; Patient Navigator services (including Informational support, Educational information, Motivational/Emotional support, Skill Building activities); Mental Health Services; and On-Site Substance Abuse Treatment (including Motivational Enhancement Therapy and Cognitive Behavioral Therapy).
  Arms: Intervention

SUMMARY:
This study will evaluate the efficacy of an integrated "Retention Clinic" in achieving virologic suppression among HIV-infected cocaine (including crack) users by using a two-group randomized, prospective trial. A total of 360 HIV-infected individuals who report cocaine (including crack) use will be randomized across study sites. The primary hypothesis is that more participants randomized to the "Retention Clinic" will have undetectable viral load than will participants randomized to the treatment as usual group.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of an integrated "Retention Clinic" in achieving virologic suppression among HIV-infected cocaine (including crack) users by using a two-group randomized, prospective trial.

Participants will be randomized to one of two groups: 1) "Retention Clinic" group and 2) Treatment as Usual. The intervention content of these groups is briefly described below:

Retention Clinic (RC) Group: This group will receive comprehensive and integrated services from a Retention Clinic. Services include HIV primary care, substance abuse treatment and mental health services, as needed. Participants in this group will also receive hands-on assistance with navigating through the clinic and accessing these services from a patient navigator.

Treatment as Usual (TAU) Group: This group will receive no protocol directed intervention. They will get the standard retention services from their local clinic.

All participants will provide informed consent and will complete a baseline audio computer-assisted self-interview or ACASI focusing on drug use, mental health, demographics and socio-economic factors, HIV care, and drug treatment history as well as blood draws for viral load and CD4 count. Follow-up assessments consisting of both ACASI and blood draws in all groups will be collected at 6 and 12 months post-randomization. Medical records will be reviewed to document use of HIV care, drug treatment and mental health services during the study period.

ELIGIBILITY:
Inclusion Criteria:

Participating individuals must:

1. be at least 18 years old
2. be HIV-seropositive (confirmed via medical record/laboratory results or via rapid HIV test in conjunction with confirmatory test or viral load)
3. meet one of the following: a) have an (*)AIDS-defining illness OR b) have a CD4 count <350 cells/uL AND a viral load >1000 copies/mL in the medical record in the past 3 months OR c) have a CD4 count <350 cells/uL AND a viral load >200 copies/mL as obtained via baseline blood draw OR d) have a clinical profile indicative of a persistently detectable HIV viral load (>200 copies/mL) attributed to non-adherence to HIV medications as per PI evaluation of the individual and/or individual's medical record
4. report (OR have evidence in the medical record of) any cocaine (including crack) use in the past 3 months OR (**)have a positive toxicology result for cocaine via the study toxicology screen
5. agree to have their blood drawn for CD4 and viral load testing
6. report living in or near either Miami, Florida (FL), or Atlanta, Georgia (GA), and be able to return for follow-up visits
7. provide locator information
8. be able to communicate in English
9. provide written informed consent
10. sign a HIPAA Authorization form/medical record release to facilitate medical record abstraction
11. be willing to go to the study clinic

(*)Site PI discretion will be used to assess whether or not the AIDS-defining illness is a good indicator of eligibility. For example, if a patient does not meet the CD4 and viral load criteria and does have an AIDS-defining illness, the Site PI will assess the AIDS-defining illness to determine whether or not the patient is a suitable candidate for the study.

(**)Per PI discretion, the urine toxicology screen may be administered as part of the screening process if the participant's self-report and/or medical record data renders him/her ineligible on the drug use criterion.

Exclusion Criteria:

Individuals will be excluded from study participation if they:

1. do not meet any one or more of the above-described inclusion criteria
2. are receiving patient navigator services for HIV care and/or substance abuse treatment
3. have significant cognitive or developmental impairment to the extent that they are unable to provide informed consent
4. are terminated via site PI decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Virologic suppression | 12 months
  To evaluate the effectiveness of the integrated "Retention Clinic" in achieving virologic suppression (defined as having an HIV-1 viral load <200 copies/mL at 6 and 12 months) among HIV-infected cocaine (including crack) users

SECONDARY OUTCOMES:
Attendance to HIV Care Visits | 12 months
  To evaluate the effectiveness of the integrated care Retention Clinic in increasing attendance at HIV care visits.
Adherence to HIV Treatment Regimens | 12 months
  To evaluate the effectiveness of the integrated care Retention Clinic in increasing adherence to HIV treatment regimens.
Attendance to Substance Abuse Treatment | 12 months
  To evaluate the effectiveness of the integrated care Retention Clinic in increasing attendance at substance abuse treatment.
Decreasing Substance Use | 12 months
  To evaluate the effectiveness of the integrated care Retention Clinic in decreasing substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R. Metsch, Ph.D., Principal Investigator — Columbia University; Carlos del Rio, M.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Jackson Health System-Special Immunology Clinic, Miami, Florida
  - Grady Health System-Ponce De Leon Center, Atlanta, Georgia

REFERENCES:
- [Derived] Metsch LR, Feaster DJ, Gooden LK, Pan Y, Parish CL, Waldrop D, Rodriguez A, Colasanti JA, Armstrong WS, Root C, Del Rio C, Castellon PC, Miller M, Pereyra MR. Project RETAIN: Providing Integrated Care for People With HIV Who Use Cocaine. Open Forum Infect Dis. 2025 Mar 3;12(4):ofaf104. doi: 10.1093/ofid/ofaf104. eCollection 2025 Apr. PMID 40276720